CLINICAL TRIAL: NCT00752336
Title: Prospective Intervention Study to Improve HRQoL and Exercise Tolerance After Heart Transplantation
Acronym: Ergo-HTx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Kugler, Christiane, PhD, Hannover Medical School, Hannover
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HTx-2777
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Exercise Capacity; Heart Transplantation
Keywords: HRQoL; exercise capacity
MeSH Terms: interventions — Exercise; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: exercise training; psychosocial support — supervised home-based endurance training; recommendation to exercise every other day

SUMMARY:
A prospective, interventional rehabilitation program was initiated to improve exercise tolerance and psychosocial functioning in patients after heart transplantation (HTx) and to evaluate long-term effects on health-related quality of life (HRQoL).Study subjects were randomized to either intervention or to control group and were followed with regular cardiopulmonary exercise testings and HRQoL measurements (SF-36) for 36±3 months after HTx. Patient characteristics did not differ concerning age, gender, and diagnosis at study entry. IG patients received regular psychosocial support and performed a home-based supervised ergometer training program. CG patients were recommended to perform regular exercising.

ELIGIBILITY:
Inclusion Criteria:

Heart transplant (6-9 mts post Tx) stabile health condition at study entry (pt stays within home environment)

* Age ≥ 18 yrs
* Sufficient language skills to answer questionnaire
* Follow-up at our center
* Willingness to participate by written informed consent

Exclusion Criteria:

* TVP diagnosis before study inclusion
* Episodes of recurrent acute rejections
* Medical contra-indication for regular exercise ergometer training
* Malignancy

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2002-01; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
HRQoL,exercise capacity | 36 mts

SECONDARY OUTCOMES:
Weight gain; cardiovascular risk factors; social re-integration | 36 mts